CLINICAL TRIAL: NCT04518982
Title: Sintilimab and Lenalidomide as a Treatment for CAEBV：a Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Sintilimab and Lenalidomide as a Treatment for CAEBV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhao Wang (Other)
Responsible Party: Sponsor-Investigator, Zhao Wang, Principal Investigator, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sintilimab,Lenalidomide,CAEBV
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: CAEBV
MeSH Terms: interventions — sintilimab; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental)
  Interventions: Drug: Sintilimab and lenalidomide
- The control group (Placebo Comparator)
  Interventions: Drug: Sintilimab placebo and lenalidomide placebo

INTERVENTIONS:
Drug: Sintilimab and lenalidomide — Drug: Sintilimab 200mg ivgtt on day 1. Drug: lenalidomide 10mg orally once a day, day 1-14.
  Arms: The experimental group
Drug: Sintilimab placebo and lenalidomide placebo — Drug: Sintilimab placebo ivgtt on day 1. Drug: lenalidomide placebo orally once a day, day 1-14.
  Arms: The control group

SUMMARY:
This study is a multi-center, prospective, randomized, controlled clinical study to evaluate the effectiveness of a combination regimen of Sintilimab and lenalidomide in patients with chronic active EBV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CAEBV confirmed by WHO criteria.
2. The Eastern United States Oncology Cooperative group (ECOG) Physical Status score is 0 or 1.
3. Before the study, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3× normal upper limit (ULN); Total bilirubin ≤2 times the normal upper limit; Serum creatinine ≤1.5 times the normal value.
4. Absolute neutrophil count ≥1×109/L; Platelet ≥50×109/L; Hemoglobin ≥60 g/L.
5. International standardized ratio ≤2.0, prothrombin time ≤1.5×ULN.
6. A woman of childbearing age must be determined not to be pregnant by a pregnancy test and is willing to take effective measures to prevent pregnancy during the trial period and ≥12 months after the last administration of the drug; All male subjects used contraceptive methods during the study period and ≥6 months after the last administration;
7. Sign the informed consent.

Exclusion Criteria:

1. There is evidence that EBV is associated with hematologic disease or malignancy, such as hemophagocytic syndrome, lymphoma-like granulomatosis, post-transplant lymphoproliferative disease, non-Hodgkin's lymphoma, Burkitt lymphoma, nasopharyngeal cancer, and gastric cancer.
2. Symptomatic EBV-associated diseases of the major organs, including the central nervous system and lungs.
3. Abnormal thyroid function.
4. Patients with grade II or above heart disease (including grade II) were identified according to the New York Heart Association (NYHA) score.
5. Have received any of the following treatments: PD-1 antibody, PD-L1 antibody or lenalidomide; Received any research drug within 12 weeks prior to the first use of the study drug; Another clinical study was also included.
6. Other primary malignancies occur within 5 years before the first administration of the drug, except those that are locally curable after radical treatment (such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma of the prostate, cervix or breast in situ, etc.).
7. A history of organ transplantation (such as liver transplantation, kidney transplantation, etc.).
8. Hematopoietic stem cell transplantation is expected during the study period.
9. Active hepatitis B (defined as hepatitis B surface antigen [HBsAg] positive during screening, or hepatitis B virus DNA titer test in peripheral blood greater than 1×103 copies/ml), and active hepatitis C (defined as hepatitis C antibody [HCV-AB] and HCV-RNA positive during screening). Serum HIV antigen or antibody positive. A history of syphilis.
10. Had major surgery within 4 weeks prior to the first medication or was expected to require major surgery during the study period.
11. Pregnant and lactating women;
12. A history of serious mental illness or drug abuse;
13. Uncontrollable infections (including lung infections, intestinal infections, etc.); Internal organ active massive hemorrhage (including gastrointestinal hemorrhage, alveolar hemorrhage, intracranial hemorrhage, etc.);
14. Allergic to the test drug ingredients or to a more severe allergic constitution;
15. Patients who cannot comply during the trial and/or follow-up phase.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | Twelve weeks after treatment
  The rate of decline in ebV-DNA copy (defined as a 2log decrease in EBV-DNA copy) or negative rate in peripheral blood mononuclear cells and plasma

SECONDARY OUTCOMES:
Spleen size | Twelve weeks after treatment
T and B lymphocyte subsets | Twelve weeks after treatment
Pathological tissue or bone marrow | Twelve weeks after treatment
treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 years
  Adverse events including thyroid function， liver function damage, myelosuppression, infection, bleeding and so on.
survival | 1 year
  From enrollment until death or the end of the experiment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No